CLINICAL TRIAL: NCT06885931
Title: Exploratory Safety and Feasibility Study of Personalized Adaptive Pudendal Neuromodulation for Mixed Urinary Incontinence and Extended Indications Using an Implanted (Picostim IITM) System
Brief Title: Augmenting Urinary Reflex Activity Study 4 (Including eXtended Indications)
Acronym: AURA-4X
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amber Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS-01529
Record Dates: First submitted 2025-03-06; First posted 2025-03-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Mixed Urinary Incontinence; Stress Urinary Incontinence (SUI); Chronic Pelvic Pain
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): Mixed Urinary Incontinence cohort
  Interventions: Device: Pudendal neuromodulation
- Cohort B (Experimental): Extended indications cohort (Stress Urinary Incontinence, Chronic Pelvic Pain, AURA-2)
  Interventions: Device: Pudendal neuromodulation

INTERVENTIONS:
Device: Pudendal neuromodulation — In this feasibility study, all subjects will receive the Amber UI system.

SUMMARY:
Exploratory safety and feasibility study of personalized adaptive pudendal neuromodulation for mixed urinary incontinence and extended indications using an implanted (Picostim™ II) system.

ELIGIBILITY:
Inclusion Criteria:

* Female. NB: the definition of female refers to sex at birth.
* Adult: aged ≥ 22 years (at the time of informed consent signature).
* Patient self-reports both stress and urge episodes (clinician-opinion on history taking).
* Patient has failed to respond to or could not tolerate conservative treatment as determined by the treating health care provider.
* Duration of urinary incontinence symptom ≥ 6 months prior to the screening baseline visit date.
* Able and willing to voluntarily sign informed consent form.
* Able to participate in all testing and follow-up clinic visits associated with study protocol.
* Patient is mobile and able to use a toilet.
* In the opinion of the Investigator, the patient is capable of independently using the system components (after training).

Exclusion Criteria:

* Patient is pregnant, breastfeeding, or plans to become pregnant at any time in the future.
* Patient is unwilling or unable to use contraception during sexual intercourse for the duration of the study.
* In the event that patient becomes pregnant during or after the study, they are not prepared to inactivate device for the whole period of the pregnancy.
* Any significant medical condition that, in the opinion of the Investigator, is likely to interfere with study procedures, device operation, or likely to confound evaluation of study endpoints.
* History of major psychiatric or personality disorder.
* Any neurological condition that in the opinion of the investigator may interfere with normal bladder function (e.g., stroke, multiple sclerosis, Parkinson's disease, clinically significant peripheral neuropathy, or complete spinal cord injury).
* Uncontrolled type I or type II diabetes (as defined by their routine care clinician or HBA1C ≥ 7.0).
* History of cancer within 5 years prior to enrolment, except for a cancer that was determined to be free of systemic cancer risk, such as basal cell carcinoma.
* Patient is taking antiplatelet and/or anticoagulant drugs including warfarin or newer alternatives (e.g., rivaroxaban, apixaban, dabigatran, edoxaban) which cannot be paused prior to surgery, or has a bleeding disorder that cannot be corrected prior to surgery.
* Any clinical reason that, in the opinion of the Investigator, may compromise patient's safety during the study.
* Currently participating in another interventional study. This excepts purely observational studies, e.g., registries.
* Patient participation in vigorous physical activities where these cannot be restricted for a period of 6 weeks post-implantation.
* Patient unwilling to stop any future participation in scuba diving below 10m. BMI ≥ 40kg/m2 or waist circumference > 106cm
* Documented history of allergic response to titanium, zirconia, polyurethane, epoxy, or silicone.
* Skin, orthopedic or neurological anatomical limitations at the site of implant that could prevent successful placement of an electrode or IPG. This includes active perineal sepsis or perianal sepsis (e.g., anal fistula and pilonidal sinus).
* Knowledge of planned MRIs, diathermy, microwave exposure, high output ultrasonic exposure, or RF energy exposure.
* Implantable neurostimulator or antennae, pacemaker or defibrillator in-situ (anywhere in body).

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 56 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Summative rates of procedural and device related adverse events and device deficiencies. | 12 months
Urinary Distress Inventory score change | 6 months
  Score minimum 0 to maximum 100. Lower score is better outcome.
Proportion of participants requiring surgical reintervention. | 12 months

SECONDARY OUTCOMES:
Urinary Distress Inventory (total, total Mixed Urinary Incontinence) score change | 12 months
  Score minimum 0 to maximum 100. Lower score is better outcome.
3-day voiding diary number of events | 12 months
  Fewer events is better outcome.
24-hour pad test weight change | 12 months
  Lower weight is better outcome.
The International Consultation on Incontinence Questionnaire score change | 12 months
  Score minimum 0 to maximum 21. Lower score is better outcome.
Patient Global Impression of Improvement score change | 12 months
  Score minimum 0 to maximum 7. Lower score is better outcome.
General Anxiety Disorder score change | 12 months
  Score minimum 0 to maximum 21. Lower score is better outcome.
Patient Health Questionnaire 9 score change | 12 months
  Score minimum 0 to maximum 27. Lower score is better outcome.
World Health Organization Disability Assessment Schedule score change | 12 months
  Score minimum 0 to maximum 100. Lower score is better outcome.
European Quality of Life 5 Dimension Questionnaire score change. | 12 months
  Score minimum 5 to maximum 25. Higher score is a better outcome.

OTHER OUTCOMES:
Numeric pain rating scale (NPRS) score change (Cohort B Chronic Pelvic Pain only) | 12 months
  Score minimum 0 to maximum 40. Lower score is better outcome.

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ghent University Hospital, Ghent
- Maastricht UMC, Maastricht, Netherlands
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No